CLINICAL TRIAL: NCT03217799
Title: Noninvasive Measurement of Blood Coagulation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, ORLY AVNERY, Senior Hematologist, Meir Medical Center
Other Study IDs: 0227
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-04

CONDITIONS: Anticoagulants; Increased; Anticoagulant Overdosage; Coagulation Disorder; Blood Clot; Blood Coagulation Disorder
MeSH Terms: conditions — Hemostatic Disorders; Thrombosis; Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Measurement of coagulability of blood — A small pneumatic cuff is attached to the root of the index finger. The sensor cuff is attached several centimeters distal to the pneumatic cuff. Measurement is taken for a 60-second control period, and then the pneumatic cuff is inflated to above-systolic blood pressure (200 mm Hg) for 180 seconds, and measurement is taken during this period of time. The cuff is then deflated, and another 60-second measurement is taken. Data is collected by the measuring device for later analysis.

SUMMARY:
The investigators have developed an optical system that measures the coagulation status of patients in vivo in a non-invasive manner. The system is based on a small optical sensor that emits coherent light into the skin and collects the reflected light from the red blood cells in the blood vessels in the skin under the sensor. The sensor is placed on the fingertip, and during a brief period of occlusion of blood flow by a small pneumatic cuff, red cell movement becomes Brownian in nature and is thereby affected by the viscosity of the blood. In patients who have a bleeding tendency, red blood cell movement will be faster, while in patients with a hypercoagulable state the red cell movement will be slower. Treatment with anticoagulant medications is expected to affect the movement of the red blood cells and these changes can be detected by the sensor. The investigators plan to test the device in normal subjects and in subjects taking Coumadin, direct oral anticoagulants, antiplatelet drugs and heparin-based medications. The investigators will determine whether anticoagulants affect the noninvasive measurement and compare the results with standard laboratory tests of coagulation.

DETAILED DESCRIPTION:
Overview: The investigators plan to measure the coagulation status with the new sensor in patients who are attending the Coagulation Clinic in Meir Hospital Center. The investigators will measure their coagulation status with the new sensor during the participants' routine clinic visits. During their visits, The participants' care will not be affected or influenced by the results of the data obtained by the new sensor. The accumulated data will be collected and later correlated with their clinical status and with routine clotting parameters that are measured, depending on the type of anticoagulation the participants receive. Specifically, in those receiving warfarin, INR will be assessed during their visit, while in patients receiving direct oral anticoagulants (DOACs), factor Xa activity will be assessed. Inparticipants receiving heparin, PTT will be assessed.

Patients and control subject: Subjects will be recruited from the Coagulation Clinic. The participants will consist of patients attending the clinic for follow-up of their prescribed anticoagulation treatment. Patients to be studied will include subjects receiving warfarin anticoagulation, NOACs, heparin and anti-platelet therapy (aspirin, clopidrogel or other anti-platelet medications). Normal subjects receiving no anticoagulation will also be studied and will serve as the control group.

Protocol: Experimental subjects will be selected from patients attending the Coagulation Clinic. Patients will be seen in the clinic and receive their usual follow-up care. After obtaining informed consent, the participants' coagulation status will be assessed with the new sensor. Patients on warfarin medications will have a venous blood sample obtained (5 ml) for determination of INR. Patients receiving NOACs will have a venous blood sample obtained (5 ml) for determination of Factor Xa activity. At a later date, the coagulation status of the patients as assessed by the new sensor will be compared to the coagulation status as assessed by the standard laboratory methods.

Normal controls will be recruited from hospital personnel. Normal controls will have their coagulation status assessed by the new sensor only. Since normal control are not receiving anticoagulation therapy, blood samples for measurement of INR or factor Xa activity will not be drawn. Normal controls will receive no financial compensation.

Methodology: The pneumatic cuff is attached to the root of the index finger. The sensor cuff is attached several centimeters distal to the pneumatic cuff. Measurement is taken for a 60-second control period, and then the pneumatic cuff is inflated to above-systolic blood pressure (200 mm Hg) for 180 seconds, and measurement is taken during this period of time. The cuff is then deflated, and another 60-second measurement is taken. Data is collected by the measuring device for later analysis.

ELIGIBILITY:
Inclusion Criteria:

Subjects receiving anticoagulant therapy, including warfarin, DOACS, heparin, and antiplatelet drugs

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending the Coagulation clinic at Meir Hospital
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of coagulability measurement with device vs. Prothrombin time | One day
  In participants taking coumadin derivatives the results of the coagulation measurement obtained with the device will be compared to results of the Prothrombin time, in seconds, and INR
Comparison of coagulability measurement with device vs. anti-Xa activity | One day
  In participants taking coumadin derivatives the results of the coagulation measurement obtained with the device will be compared to results of the anti-Xa activity, measured as anti-Xa units/ml
Comparison of coagulability measurement with device vs. PTT | one day
  In participants taking heparin the results of the coagulation measurement obtained with the device will be compared to results of the PTT, seconds

IPD SHARING:
Plan to Share IPD: No